CLINICAL TRIAL: NCT07113431
Title: A Novel Partial-enteral Nutrition Protocol to Improve Nutrition Status of Adults Patients Experiencing a Crohn's Disease Flare and Starting New Immunologic Therapy.
Brief Title: Partial-enteral Nutrition Protocol for Crohn's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kate Farms Inc (Industry)
Collaborators: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UMN2023
Record Dates: First submitted 2025-07-24; First posted 2025-08-08 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Crohn's Disease(CD)

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IBD-AID diet (Placebo Comparator)
  Interventions: Other: IBD-AID diet
- IBD-AID Diet + Kate Farms Peptide 1.5 (Active Comparator)
  Interventions: Dietary Supplement: IBD-AID diet combined with Kate Farms Peptide 1.5

INTERVENTIONS:
Dietary Supplement: IBD-AID diet combined with Kate Farms Peptide 1.5 — Combining standardized-IBD diet developed by the University of Minnesota (IBD-AID) with commercially available pea protein plant-based enteral nutrition formula (Kate Farms Peptide 1.5)
  Arms: IBD-AID Diet + Kate Farms Peptide 1.5
Other: IBD-AID diet — Standardized IBD diet developed by the University of Massachusetts Medical School (IBD-AID)
  Arms: IBD-AID diet

SUMMARY:
A novel dietary intervention combining a standardized IBD diet (IBD-AID) with supplementation from a pea protein plant-based oral nutrition supplement (ONS) (Kate Farms Peptide 1.5) to improve protein, calorie, and nutrient intake in adult patients experiencing a Crohn's disease flare starting new immunologic therapy. Additionally, this study will include objective measures of body composition to improve nutrition status assessment and provide a more sensitive measure of intervention efficacy compared to anthropometric measures of body weight or BMI.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe CD as defined by physician and starting new biologic therapy
* Able and willing to complete the study procedures
* Age > 18
* Able to comply with study measures in the opinion of the investigator

Exclusion Criteria:

* Diagnosis of short bowel syndrome
* Presence of ileostomy or colostomy
* Presence of a pacemaker or any electronic implantable device
* Use of pre or probiotic supplements within 14 days of randomization
* High risk for development of refeeding syndrome
* In the opinion of the investigator would not complete the study procedures
* Patients with active implanted medical devices, e.g. cardiac pacemakers, defibrillators or patients connected to electronic life support devices
* Pregnant Patients: while the use of bioimpedance technology in pregnant patients has been shown to have no adverse effects, it has yet to be clinically validated for use with that population group
* Serious, concomitant illness that, in the opinion of the investigator would interfere with evaluation of safety or efficacy, or put the participant at risk of harm from study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2025-10-24 (Actual); Study Completion 2025-10-24 (Actual)

PRIMARY OUTCOMES:
Nutrient intake | 8 weeks
  Nutrient intake improvement assessed by 24-hour dietary recall from a combined intervention of a standard IBD-AID diet with an oral nutrition supplement drink (Kate Farms Peptide 1.5) compared to a standard diet alone without an oral nutrition supplement drink.

SECONDARY OUTCOMES:
Body composition | 8 weeks
  Body composition measures assessed by bioimpedance spectroscopy (BIS).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Undecided